CLINICAL TRIAL: NCT06484894
Title: The Effect of Refractive Errors on Central Corneal Thickness by Using Pentacam
Brief Title: The Effect of Refractive Errors on Central Corneal Thickness by Using Pentacam and IOL Master
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidy Nayer Adly, Resident doctor, Assiut University
Other Study IDs: Central corneal thickness
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Central Corneal Thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypermetrope: Effect of hypermetropia on central corneal thickness by using pentacam and IOL master
  Interventions: Device: Pentacam and IOL master
- Emmetrope: Effect of emmetropia on central corneal thickness by using pentacam and IOL master
  Interventions: Device: Pentacam and IOL master
- Myopia: Effect of myopia on central corneal thickness by using pentacam and IOL master
  Interventions: Device: Pentacam and IOL master

INTERVENTIONS:
Device: Pentacam and IOL master — Device used for measurement of central corneal thickness

SUMMARY:
To evaluate the impact of refractive errors on the central corneal thickness obtained by Pentacam and intraocular lenses (IOL) master in eyes with different refractive errors.

DETAILED DESCRIPTION:
Central corneal thickness (CCT) is a key indicator of corneal health status and helps to assess corneal diseases. The normal corneal thickness is about 540 μm and mainly consists of the stroma, which is estimated at 450 μm in the center. The stroma provides vital structural integrity and plays a key role in helping maintain transparency. It has been reported, however, that CCT follows a diurnal pattern being 10 μm thicker in the morning due to reduced evaporation of water from underneath the closed eyelids

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in this study aged between20 and 41 years, asked for refractive surgery

Exclusion Criteria:

* patients with corneal scarrig or opacification.

  * Patients with corneal dystrophies.
  * Patients with keratoconus.
  * Previous ocular or refractive surgery.
  * Ocular trauma.
  * Uveitis patients.
  * Patients with history of recent contact lens wear.

Ages: 20 Years to 41 Years | Sex: All
Age Groups: Adult
Study Population: 1. Inclusion criteria:
     Subjects included in this study aged between20 and 41 asked for refractive surgery
  2. Exclusion criteria:-
     * Severe corneal scarrig or opacification., dystrophy
     * Patients with history of recent contact lens Ocular trauma.
     * Uveitis patients Patients with keratoconus.
     * Previous ocular or refractive surgey
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To find if there a correlation between refractive errors and the central corneal thickness | Baseline
  Study the effect of refractive errors on central corneal thickness

SECONDARY OUTCOMES:
To study if there a difference between measurement by pentacam and measurement of IOL master | Baseline
  Study which device is more accurate in measuring the central corneal thickness and if there is any difference between the two devices

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Fathy rateb, Professor, Study Director — Assiut University; Ahmed Abd el Nasser awad, Lecturer, Study Chair — Assiut University; Mohamed Tarek Abd el menaam, Professor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Wang Q, Liu W, Wu Y, Ma Y, Zhao G. Central corneal thickness and its relationship to ocular parameters in young adult myopic eyes. Clin Exp Optom. 2017 May;100(3):250-254. doi: 10.1111/cxo.12485. Epub 2016 Oct 18. PMID 27757993
- [Background] Prasad A, Fry K, Hersh PS. Relationship of age and refraction to central corneal thickness. Cornea. 2011 May;30(5):553-5. doi: 10.1097/ICO.0b013e3181fb880c. PMID 21107245